CLINICAL TRIAL: NCT01659359
Title: Vice-presidency for Research
Brief Title: The Effect of Virtual Reality Glasses on Pain and Anxiety
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Samira Ebrahimzadeh Zagami, Principle Investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: virtual reality glasses
Record Dates: First submitted 2012-08-04; First posted 2012-08-07 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Pain and Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- virtual reality glasses and Lidocaine (Experimental): virtual reality glasses and 5 ml Lidocaine 2%
  Interventions: Device: Virtual reality glasses and Lidocaine
- Lidocaine (Experimental): 5 cc Lidocaine2%
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Device: Virtual reality glasses and Lidocaine — The samples were randomly allocated to use Virtual reality glasses and 5 ml Lidocaine2% for decreasing pain and anxiety in episiotomy repair.
  Arms: virtual reality glasses and Lidocaine
Drug: Lidocaine — The samples were randomly allocated to use 5 ml Lidocaine2% for decreasing pain and anxiety in episiotomy repair.
  Arms: Lidocaine

SUMMARY:
In recent studies using virtual reality has been proposed as a non pharmacological methods for pain relief but until this time , its effects has not been assessed on pain and anxiety during episiotomy repair. To determine the effectiveness of virtual reality Glasses on pain and anxiety in Primiparity women during episiotomy repair.

ELIGIBILITY:
Inclusion Criteria:

* Iranian
* low risk pregnancy
* Apgar ≥ 7

Exclusion Criteria:

* vision or ear disorders
* History of motion sickness or headaches
* psychological disease or Addiction
* Prescribe narcotic or sedation 4hour prior to delivery.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Virtual reality glasses decreased pain and anxiety during episiotomy | up to 8 months